CLINICAL TRIAL: NCT05505474
Title: Use of a Subcutaneous Catheter for Controlled Ovarian Stimulation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Southern California (Other)
Collaborators: ConvaTec Inc. (Industry)
Responsible Party: Principal Investigator, Richard Paulson, Professor, University of Southern California
Other Study IDs: APP-21-05650
Record Dates: First submitted 2022-05-19; First posted 2022-08-17 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- IVF with Neria™ Guard device: Patients undergoing IVF with the use of the Neria™ Guard subcutaneous catheter
  Interventions: Device: IVF with the Neria™ Guard Subcutaneous Catheter

INTERVENTIONS:
Device: IVF with the Neria™ Guard Subcutaneous Catheter — Use of the Neria™ Guard subcutaneous catheter for administration of subcutaneous medication in an IVF cycle.

SUMMARY:
Subcutaneous medications are an integral part of controlled ovarian stimulation protocols for in-vitro fertilization (IVF), but daily or twice daily injections are both physically and emotionally burdensome for patients and their partners. This is a feasibility study to evaluate the use of the Neria Guard™ (Unomedical, Convatec) subcutaneous catheter for ovarian stimulation in IVF.

DETAILED DESCRIPTION:
Daily or twice daily injections are a standard part of controlled ovarian stimulation for in-vitro fertilization (IVF). These injections are both physically and emotionally burdensome for patients and contribute additional stressors to those already inherent to infertility. Subcutaneous catheters have been demonstrated to be effective for administration of insulin, anticoagulants, and other medications in pediatric patients, and subcutaneous gonadotropin-releasing hormone pumps have also been used in hypothalamic patients. This study aims to assess the feasibility of a subcutaneous catheter in patients undergoing ovarian stimulation for IVF. Primary outcomes will include the incidence of safety and catheter-related issues as well as assessment of patient satisfaction in cycles using the subcutaneous catheter. We will also closely monitor estradiol and follicle-stimulating hormone levels during stimulation to ensure adequate medication administration via the catheter as well as IVF outcomes including mature oocyte yield, embryo maturation, and pregnancy rates.

ELIGIBILITY:
Inclusion Criteria:

* Female between 18 and 45 years of age undergoing controlled ovarian stimulation

Exclusion Criteria:

* none

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 100 patients undergoing controlled ovarian stimulation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Device feasibility | During ovarian stimulation (usually 9-12 days)
  To measure follicle-stimulating hormone (FSH) and estradiol levels after administration of subcutaneous gonadotropins via the catheter

SECONDARY OUTCOMES:
Adverse effects related to the subcutaneous catheter | During ovarian stimulation (usually 9-12 days)
  Catheter malfunction, number of times needed to administer traditional needle injection, need for premature catheter exchange or removal, emergency pages to the clinic for catheter-related issues, local issue reactions, pain, bleeding, hematoma, infection
Patient satisfaction and acceptability | During ovarian stimulation (usually 9-12 days)
  Patient satisfaction will be evaluated via a self-designed pre- and post-cycle questionnaire to quantify pre-cycle needle phobia, satisfaction with the catheter system, reasons for continuation or discontinuation. The questionnaires will be preapproved by the University of California Institutional Review Board.
Number of mature oocytes retrieved | Immediately following ovarian stimulation and oocyte retrieval
  The number of oocytes in metaphase II retrieved at the time of oocyte retrieval
Embryo blastulation | 5-7 days after oocyte retrieval
  The number of embryos that progress to blastocyst per the number fertilized
Clinical pregnancy | 1-2 weeks following embryo transfer
  As defined by a intrauterine gestational sac between weeks 5 and 6

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Paulson, MD, Principal Investigator — University of Southern California
Locations (1):
- HRC Fertility, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to publish and share deidentified data of primary and secondary outcomes.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Haemmerli Keller K, Alder G, Loewer L, Faeh M, Rohner S, von Wolff M. Treatment-related psychological stress in different in vitro fertilization therapies with and without gonadotropin stimulation. Acta Obstet Gynecol Scand. 2018 Mar;97(3):269-276. doi: 10.1111/aogs.13281. Epub 2018 Jan 8. PMID 29247514
- [Background] Burdick P, Cooper S, Horner B, Cobry E, McFann K, Chase HP. Use of a subcutaneous injection port to improve glycemic control in children with type 1 diabetes. Pediatr Diabetes. 2009 Apr;10(2):116-9. doi: 10.1111/j.1399-5448.2008.00449.x. Epub 2009 Jan 7. PMID 19175512
- [Background] de Jong ME, Carbiere T, van den Heuvel-Eibrink MM. The use of an insuflon device for the administration of G-CSF in pediatric cancer patients. Support Care Cancer. 2006 Jan;14(1):98-100. doi: 10.1007/s00520-005-0872-x. Epub 2005 Aug 12. PMID 16096770
- [Background] Hanas SR, Carlsson S, Frid A, Ludvigsson J. Unchanged insulin absorption after 4 days' use of subcutaneous indwelling catheters for insulin injections. Diabetes Care. 1997 Apr;20(4):487-90. doi: 10.2337/diacare.20.4.487. PMID 9096966
- [Background] Solnica A, Oh C, Cho MM, Loughlin JS, McCulloh DH, McGovern PG. Patient satisfaction and clinical outcome after injecting gonadotropins with use of a needle-free carbon dioxide injection system for controlled ovarian hyperstimulation for in vitro fertilization. Fertil Steril. 2009 Oct;92(4):1369-1371. doi: 10.1016/j.fertnstert.2009.03.013. Epub 2009 Apr 7. PMID 19356750